CLINICAL TRIAL: NCT07296159
Title: A Technology-enhanced and Multilevel Approach to Promote Cervical Cancer Prevention Among Women Living With HIV
Brief Title: My Self-Sampling for HPV Awareness, Results, and Empowerment
Acronym: MySHARE+
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daisy Le (Other)
Responsible Party: Sponsor-Investigator, Daisy Le, PI, George Washington University
Organization: George Washington University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5K01CA276624 (NIH)
Record Dates: First submitted 2025-12-18; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer; Cervical Cancer Screening; HPV
Keywords: Cervical cancer; HPV; HPV self-sampling; mHealth
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MySHARE+ Intervention (Experimental): Participants will receive mHealth education via automated text messages.
  Interventions: Other: MySHARE+ mHealth Education Intervention
- Control (No Intervention): Participants will received a text message welcoming them to the project with a referral link to the NCI's cervical cancer screening website with monthly reminders over the span of six months.
- Healthcare provider prompt (Other): Support with the development and refinement of provider prompt to improve communication about cervical cancer screening.
  Interventions: Other: Healthcare Provider Prompt

INTERVENTIONS:
Other: MySHARE+ mHealth Education Intervention — Participants in the intervention group will receive detailed pre-tested educational theory-based SMS messaging and education over the course of four weeks.
  Arms: MySHARE+ Intervention
Other: Healthcare Provider Prompt — Providers of healthcare and/or social services to WLH will complete an online survey to identify barriers to implementing an healthcare provider prompt in a primary care setting and participate in semi-structured interviews to provide feedback on drafted prompts. Prompts will be piloted at one local clinic to improve patient-provider communication about cervical cancer screening, followed with semi-structured interviews with providers involved.
  Arms: Healthcare provider prompt

SUMMARY:
The overall objective of this study is to conduct formative research and pilot test the provider-level and patient-level components of the My Self-Sampling for HPV Awareness, Results, and Empowerment (MySHARE+) intervention. MySHARE+ aims to harness the power of technology and apply a multilevel approach to promote the adoption of cervical cancer screening (HPV self-sampling; Pap triage adherence) among under/never-screened women living with HIV (WLH). The specific aims are to 1) identify facilitators and barriers to implementing a healthcare provider prompt in a primary care setting and 2) conduct a pilot randomized controlled trial (RCT) to examine the feasibility, acceptability, and preliminary efficacy of a mHealth educational intervention in promoting cervical cancer awareness and HPV self-sampling among WLH.

Under aim 1: Providers of healthcare and/or social services to WLH will complete an online survey to identify barriers to implementing a healthcare provider prompt in a primary care setting and participate in semi-structured interviews to provide feedback on drafted prompts. Prompts will be piloted at one local clinic to improve patient-provider communication about cervical cancer screening, followed with semi-structured interviews with providers involved.

Under aim 2: Participants will be enrolled in a text messaging intervention and sent an HPV self-sampling test kit to return via mail. Participants in the intervention group will receive the full mHealth intervention while the control group will receive more generic text messages and reminders over the course of the study.

ELIGIBILITY:
Aim 1 Provider Prompt: Healthcare and/or service provider to women living with HIV

Aim 2 RCT Pilot

Inclusion Criteria:

* Have an HIV diagnosis
* Are between 30 to 65 years old
* Have not had a Pap smear within the last 12 months or more.

Exclusion Criteria:

* Have had a history of hysterectomy or invasive cervical cancer
* Are currently pregnant or were pregnant in the past 3 months
* Are currently participating or enrolled in similar studies within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who received and used the mailed HPV self-sampling kit. | 1 month, 3 months, and 6 months
  Feasibility of the mailed HPV self-sampling program: number of participants who received and used the HPV self-sampling test over the number of enrolled participants.
Proportion of participants who reported the presence of technical issues with the MySHARE+ messages. | 1 month, 3 months, and 6 months
  Feasibility of the MySHARE+ text-messaging program: number of participants who reported technical issues over the number of enrolled participants.
Proportion of participants who received all text messages and engaged with the MySHARE+ educational program. | 6 months
  Feasibility of the MySHARE+ text-messaging program: number of participants who received and engaged with 100% of the MySHARE+ messages over the number of participants enrolled in the text-messaging program.
Proportion of participants who were satisfied with the HPV self-sampling test. | 1 month, 3 months, and 6 months
  Acceptability of the HPV self-sampling test: number of participants satisfied with the HPV self-sampling test (e.g., understanding of instructions, ease of use, degree of pain and bleeding associated with use, and willingness to use self-sample HPV testing regularly using a 5-point Likert scale) over the number of enrolled participants.
Proportion of participants who were satisfied with the MySHARE+ text-messaging program | 1 month, 3 months, and 6 months
  Acceptability of the MySHARE+ text messaging program: number of participants with rated satisfaction items as four or higher from a 5-point Likert scale over the number of enrolled participants.
Proportion of participants who unsubscribed from the MySHARE+ text-messaging program. | 1 month, 3 months, and 6 months
  Acceptability of the MySHARE+ text messaging program: number of participants who unsubscribed from the MySHARE+ text-messaging program over the number of enrolled participants. An unsubscription rate of 15% or less will be considered acceptable
Proportion of participants who returned the HPV self-sampling test within three months of enrollment. | 1 month, 3 months
  Preliminary efficacy of the HPV self-sampling and the MySHARE+ mHealth program: number of participants who returned the HPV self-sampling test within three months of enrollment over the number of enrolled participants.

SECONDARY OUTCOMES:
Proportion of participants who completed an in-clinic follow-up Pap test since baseline. | 1 month, 3 months, and 6 months
  Preliminary efficacy of the HPV self-sampling and the MySHARE+ mHealth program: number of participants who completed an in-clinic Pap test over the number of enrolled participants.
Proportion of participants with an HPV positive test who completed an in-clinic follow-up Pap test since baseline. | 1 month, 3 months, and 6 months
  Preliminary efficacy of the HPV self-sampling and the MySHARE+ mHealth program: number of participants with an HPV positive test who completed an in-clinic Pap test over the number of participants with an HPV+ test.

IPD SHARING:
Plan to Share IPD: No